CLINICAL TRIAL: NCT02918006
Title: Phase 2 Randomized, Controlled, Human Influenza A (H1N1) Challenge Study Following Administration of an Oral H1N1 HA Adenoviral-Vector Based Seasonal Influenza Vaccine and dsRNA Adjuvant to Healthy Adult Volunteers
Brief Title: A Phase 2 Influenza A Challenge Study Following Oral Administration of an H1N1 HA Ad-Vector Seasonal Flu Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxart (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA-CHAL-201
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Influenza
Keywords: Challenge; oral vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Oral vaccination followed by viral challenge at 3 months post vaccination
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Vaccine (VXA-A1.1) (Experimental): Oral enteric coated vaccine tablets. Placebo (saline solution) IM injection will also be administered in this arm.
  Interventions: Biological: VXA-A1.1; Other: Saline Solution for Placebo IM Injection
- QIV IM Injection (Active Comparator): A commercially available QIV will be administered at the approved dose level as the active comparator. Oral placebo tablets will also be administered in this arm.
  Interventions: Biological: Fluzone®; Other: Placebo Tablets
- Oral and IM Placebo (Placebo Comparator): Two forms or placebos (saline IM injection and oral placebo tablets) will be administered in this arm.
  Interventions: Other: Placebo Tablets; Other: Saline Solution for Placebo IM Injection

INTERVENTIONS:
Biological: VXA-A1.1 — Enteric coated oral vaccine tablet
  Other Names: Oral H1N1 Ad5 Tableted Vaccine
  Arms: Oral Vaccine (VXA-A1.1)
Biological: Fluzone® — Fluzone Quadravalent (Fluzone®) influenza vaccine (QIV) suspension for intramuscular (IM) injection
  Other Names: Fluzone Quadravalent
  Arms: QIV IM Injection
Other: Placebo Tablets — Placebo tablets similar in size, color and number to the active oral tablet vaccine drug product
  Other Names: Enteric Coated Placebo Tablets
  Arms: Oral and IM Placebo; QIV IM Injection
Other: Saline Solution for Placebo IM Injection
  Other Names: 0.9% Sodium Chloride Injection, USP
  Arms: Oral Vaccine (VXA-A1.1); Oral and IM Placebo

SUMMARY:
A Phase 2 Randomized, Placebo- and Active-Controlled, Human Influenza A/California/04/2009 (H1N1) Challenge Study Following Administration of an Oral H1N1 Hemagglutinin (HA) Adenoviral-Vector Based Seasonal Influenza Vaccine and dsRNA Adjuvant (VXA-A1.1) to Healthy Adult Volunteers.

DETAILED DESCRIPTION:
This is a Phase 2 randomized, placebo- and active-controlled, two-part study in which healthy adult volunteers with low or undetectable pre-existing antibodies against A/California/7/2009(H1N1) pdm09-like virus will be challenged with an influenza A/H1N1 human challenge strain approximately 90 days after vaccination with a single dose of H1N1 HA Adenoviral-vector based seasonal influenza vaccine and dsRNA adjuvant (VXA-A1.1), an injectable QIV vaccine, and/or placebo.

An independent Safety Monitoring Committee (SMC) will oversee the safety of the study.

To accommodate the limited size of the isolation unit that will be utilized for the challenge and post-challenge sequestration period, subjects will move through the study (enrollment, vaccination and challenge) sequentially in a total of 6 cohorts. Each cohort will randomize 30 subjects to obtain approximately 25 subjects per cohort for the challenge phase. Subjects will be randomized in a ratio of 2:2:1 (VXA-A1.1: Quadrivalent Influenza Vaccine (QIV): Placebo.

The study will be conducted in two parts.

Part A: Subjects will be randomized in a double-blinded manner to receive a single administration of one of three treatment arms:

* Arm 1: VXA-A1.1 oral vaccine + placebo Intramuscular (IM)
* Arm 2: QIV (IM) injection + oral placebo
* Arm 3: Placebo IM injection + oral placebo

Subjects will return to the site for ~8 visits and be contacted remotely at defined time points to be followed for immunogenicity and safety during study Part A.

Part B: Subjects will be challenged with a wild-type influenza A H1 virus strain ~90 days following vaccination. Blood samples will be collected to evaluate immunogenicity. Subjects will remain in the isolation unit for 6 to 9 days post-challenge.

Following challenge, influenza symptoms and signs will be assessed during the sequestration period. Blood samples and nasopharyngeal swab samples will be collected. Vital signs will be measured every 4 hours during waking hours.

After release from the isolation unit subjects will return to the site 30 days post-challenge. Part B will continue for purposes of collecting long term safety follow-up (serious adverse events (SAEs), AEs of special interest (AESIs) and any new onset of chronic illness (NOCI) via phone contacts through 1 year post-vaccination (Day 365).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18 - 49 years, inclusive
2. Able to give written informed consent
3. Low pre-existing antibodies to the study vaccine
4. In general good health (no clinically significant health concerns)
5. Safety laboratory normal range or not clinically significant (NCS), with few exceptions
6. Body mass index (BMI) between 17 and 35
7. Comprehension of the study requirements with ability and willingness to complete all assessments and comply with scheduled visits and contacts
8. Female participants must have a negative pregnancy test at screening

Exclusion Criteria:

1. Receipt of any influenza vaccine within two years prior to study
2. Use of any investigational vaccine/adjuvanted vaccine within 8 weeks of study
3. Use of any investigational drug or device within 4 weeks of study
4. Use of any licensed vaccine within 30 days of study
5. Presence of significant uncontrolled medical or psychiatric illness within 3 months of study
6. Clinically significant and/or protocol defined ECG abnormality
7. Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies
8. Cancer, or treatment for cancer, within 3 years of study
9. History of drug, alcohol or chemical abuse within 1 year
10. Receipt of blood or blood products within 6 months of study
11. Donation of blood within 4 weeks of study
12. Presence of a fever ≥ 38ºC measured orally at baseline
13. Stool sample with occult blood at screening
14. Positive urine drug screen for drugs of abuse at screening
15. Positive breath or urine alcohol test at screening or baseline
16. Consistent/habitual smoking within 2 months prior to vaccination
17. History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, Guillain-Barre syndrome, hives or abdominal pain
18. Asthma, bronchiectasis or chronic obstructive pulmonary disease
19. Any known allergy or intolerance to oseltamivir

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Tucker, PhD, Study Director — Vaxart, Inc.
Locations (1):
- WCCT Global, Costa Mesa, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liebowitz D, Gottlieb K, Kolhatkar NS, Garg SJ, Asher JM, Nazareno J, Kim K, McIlwain DR, Tucker SN. Efficacy, immunogenicity, and safety of an oral influenza vaccine: a placebo-controlled and active-controlled phase 2 human challenge study. Lancet Infect Dis. 2020 Apr;20(4):435-444. doi: 10.1016/S1473-3099(19)30584-5. Epub 2020 Jan 21. PMID 31978354
- [Derived] McIlwain DR, Chen H, Apkarian M, Affrime M, Bock B, Kim K, Mukherjee N, Nolan GP, McNeal MM. Performance of BioFire array or QuickVue influenza A + B test versus a validation qPCR assay for detection of influenza A during a volunteer A/California/2009/H1N1 challenge study. Virol J. 2021 Feb 25;18(1):45. doi: 10.1186/s12985-021-01516-0. PMID 33632249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Aug 31, 2016, and Jan 23, 2017, 374 individuals were assessed for eligibility.
Groups:
- Oral Vaccine (VXA-A1.1): Oral enteric coated vaccine tablets. Placebo (saline solution) IM injection was also administered in this arm.
  VXA-A1.1: Enteric coated oral vaccine tablet
  Saline Solution for Placebo IM Injection
- QIV IM Injection: A commercially available QIV was administered at the approved dose level as the active comparator. Oral placebo tablets were also administered in this arm.
  Fluzone®: Fluzone Quadravalent (Fluzone®) influenza vaccine (QIV) suspension for intramuscular (IM) injection
  Placebo Tablets: Placebo tablets similar in size, color and number to the active oral tablet vaccine drug product
- Oral and IM Placebo: Two forms of placebo (saline IM injection and oral placebo tablets) were administered in this arm.
  Placebo Tablets: Placebo tablets similar in size, color and number to the active oral tablet vaccine drug product
  Saline Solution for Placebo IM Injection
Period: Allocation and Follow-Up
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo
Started | 71 | 72 | 36
Completed | 69 | 70 | 35
Not Completed | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Vaccination Phase Analysis
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo
Started | 69 | 70 | 35
Completed | 58 | 54 | 31
Not Completed | 11 | 16 | 4
Not completed — Withdrawal by Subject | 3 | 7 | 2
Not completed — Biofire Positive | 5 | 5 | 0
Not completed — Symptoms of Sinusitis | 1 | 0 | 0
Not completed — Exlcuded by Investigator for Safety of Compliance | 2 | 3 | 2
Not completed — Seasonal allergies | 0 | 1 | 0
Period: Challenge Phase Analysis
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo
Started | 58 | 54 | 31
Completed | 58 | 54 | 29
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo | Total
Number analyzed (Participants) | 71 | 72 | 36 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 72 | 36 | 179
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 15 | 73
  Male | 42 | 43 | 21 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 21 | 10 | 55
  Not Hispanic or Latino | 47 | 48 | 26 | 121
  Unknown or Not Reported | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 8 | 8 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 14 | 16 | 7 | 37
  White | 45 | 45 | 24 | 114
  More than one race | 3 | 3 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Hemagglutination Inhibition (HAI) Titer [Number; unit: participants] — Participants with a baseline HAI Titer of less than 20 were eligible for study participation.
  participants | 54 | 49 | 29 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Influenza-like Clinical Illness and Laboratory Confirmed Infection Post Challenge With a Homologous A Strain Influenza Virus
Description: The clinical efficacy of VXA-A1.1 to protect against illness caused by the homologous A strain influenza virus with challenge 3 months following a single immunization in comparison to placebo and QIV. Participants were evaluated for clinical signs and symptoms of influenza as well as for viral shedding via PCR for confirmation of infection.
Time Frame: Clinical Illness and/or laboratory confirmed infection occurring following viral challenge at 3 months post vaccination
Population: Subjects that did not complete the vaccination phase per protocol criteria, did not undergo viral challenge, did not have Biofire results positive for infections other than influenza or were discharged early from the isolation unit post challenge were excluded from the per protocol analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo
Number analyzed (Participants) | 58 | 54 | 31
Participants | 17 | 19 | 15

ADVERSE EVENTS:
Time Frame: Systemic and local solicited adverse events were collected daily through Day 8 post-vaccination Unsolicited AEs were recorded through 120 days post-vaccination (90 days in Part A and 30 days post challenge in Part B) SAEs and AESIs/NOCIs are recorded through Day 365
Description: Systemic and local solicited adverse events were graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe) Systemic events include: diarrhea, nausea, vomiting, abdominal pain, malaise, anorexia, headache, myalgia and fever. Local events include injection site reactions of: pain, tenderness, erythema, and induration.
Arm/Group | Oral Vaccine (VXA-A1.1) | QIV IM Injection | Oral and IM Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/72 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/36
Other Adverse Events (participants affected / at risk) | 15/71 | 11/72 | 4/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Vaccine (VXA-A1.1) (N=71) | QIV IM Injection (N=72) | Oral and IM Placebo (N=36)
Upper Respiratory Infection (Infections and infestations) | 11 | 7 (7) | 4
Headache (Endocrine disorders) | 4 (4) | 4 (4) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02918006/Prot_SAP_000.pdf